CLINICAL TRIAL: NCT06703255
Title: A Phase IIa Clinical Study of HX301 Alone or in Combination with Temozolomide in Patients with High-Grade Glioma (Grade III and IV)
Brief Title: A Phase 2 Study of HX301 in Patients with High-grade Giloma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hangzhou Hanx Biopharmaceuticals, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HX301-II-01
Record Dates: First submitted 2024-11-21; First posted 2024-11-25 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Patients received HX301/+Temozolomide treatment at assigned dose level on a 4 weeks basis (Experimental)
  Interventions: Drug: HX301+/Temozolomide

INTERVENTIONS:
Drug: HX301+/Temozolomide — Part I: It is planned to firstly explore a dose of 160 mg and enroll approximately 3-6 subjects to receive HX301 monotherapy until disease progression, intolerable toxicity, or other reasons for stopping treatment for up to 24 cycles of 28 days each. Safety evaluation was performed using the traditional "3 + 3" rule, and the DLT observation period was 28 days (C1D1 ~ C1D28). If 160 mg was not tolerated, it was reduced to 120 mg for exploration. Part II: Combination therapy phase: HX301 will be administered in combination with temozolomide approximately 4-6 weeks after completion of chemoradiotherapy. The TMZ dose will follow the first cycle: 150 mg/m 2 qd D1-D5, starting with the second cycle, and if the criteria for TMZ dose increase are met, TMZ will be administered as 200 mg/m 2 qd D1-D5 every 2 8 days for up to 12 cycles. Monotherapy maintain period: Following the end of temozolomide treatment, HX301 monotherapy will be continued for a maximum of 12 cycles of 28 days each.

SUMMARY:
The study will include a dose-escalation and dose-expansion component to establish the recommended Phase 2 dose (RP2D) for HX301 in combination with Temozolomide and to evaluate the preliminary antitumor activity of HX301.HX301 is an investigational drug that has not yet been approved by the Food and Drug Administration (FDA) or any other regulatory authorities for commercial purposes.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form;
2. Age ≥ 18 years;
3. Expected survival ≥ 12 weeks;
4. Part I:1) Histologically confirmed high-grade glioma (WHO classification grade III or IV); 2) At least one prior temozolomide treatment; 3) Patients with recurrent or progressive clinically assessed disease according to RANO criteria with evaluable lesions; Part II: Patients with histological or cytological diagnosis of glioblastoma according to World Health Organization (WHO) classification (2021) who received surgical treatment for the first time and standard concurrent chemoradiotherapy and who have not received any other prior treatment;
5. Part II: Subjects must undergo partial or complete surgical resection, and available results of postoperative brain contrast-enhanced MRI were documented as follows: 1) complete resection without gadolinium enhancement ; or 2) complete resection (80% or more);
6. Part II: Subjects must complete initial radiotherapy combined with TMZ (concurrent chemoradiotherapy) for glioblastoma according to the Stupp regimen (Stupp 2005) (total radiation dose 5 4-60 G y);
7. Part I: If radiotherapy has been performed, the completion of radiotherapy shall last for 3 months, or there shall be tumor progression or histopathological confirmation of progression in the original radiation field within 3 months; Part II: there shall be no evidence of disease progression after chemoradiotherapy, except for pseudo progression;
8. Dexamethasone was administered at ≤ 5 mg/day at study entry.Corticosteroids should be reduced as far as possible to the smallest dose necessary to control neurological symptoms before receiving study treatment;
9. Karnofsky performance status (KPS) ≥ 70 within 1 4days prior to receiving study treatment ;
10. Willing and able to comply with the protocol.

Exclusion Criteria:

1. Part II: Patients with recurrent glioblastoma;
2. Distant metastasis involving brainstem and meninges or extension of lesions to spinal cord;
3. Human immunodeficiency virus (HIV) antibody positive, syphilis antibody (Anti-TP) positive, hepatitis C virus (HCV) antibody positive and HCV RNA positive, hepatitis B virus surface antigen (HBsAg) positive and HBV DNA positive (HBsAg positive requires further detection of HBV DNA, HBV DNA ≥ 200 IU/ml, or ≥ 10 3 copies/ml);
4. Hypersensitivity to temozolomide and/or components of HX301;
5. At risk for torsades de pointes (TdP): patients with a marked prolongation of the QT/QTc interval calculated using the Fredericia QT correction formula at baseline (eg, repeated demonstration of QTc interval > 470 ms), or a history of other TdP risk factors (eg, heart failure, hypokalemia, family history of long QT syndrome), or patients who are currently taking medications that prolong the QT/QTc interval;
6. Grade ≥ 2 diarrhea at baseline;
7. Participation in another study involving an investigational drug within 30 days prior to the first dose of study drug;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-01-08 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Part I: Number of participants experiencing Adverse Events (AEs) | All AEs up to 28(±7)days after the last dose of study treatment
  An AE is any untoward medical occurence in a patient or subject, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Part I: Identify the recommended phase IIa dose (RP2D) of HX301 in patients with high-grade glioma; | 24 Cycles of 28 days each.
  RP2D is Recommended Phase II Dose.
Part II (HX301 monotherapy safety run-in period) : Number of participants experiencing Adverse Events (AEs) | All AEs up to 28(±7)days after the last dose of study treatment
  An AE is any untoward medical occurence in a patient or subject, temporally associated with the use of study treatment, whether or not considered related to the study treatment.
Part II (HX301 monotherapy safety run-in period) : Identify the recommended phase IIa dose (RP2D) of HX301 combination with TMZ in patients with high-grade glioma; | 24 Cycles of 28 days each.
  RP2D is Recommended Phase II Dose.
Part II (HX301 in combination with temozolomide) : Progression-free survival（PFS） per Investigator assessed using RANO criteria. | 24 Cycles of 28 days each.
Part II (HX301 in combination with temozolomide) :Objective response rate（ORR） per Investigator assessed using RANO criteria. | 24 Cycles of 28 days each.

SECONDARY OUTCOMES:
Part I : Objective response rate（ORR） per Investigator assessed using RANO criteria. | 24 Cycles of 28 days each.
Part II (HX301 monotherapy safety run-in period) : Objective response rate（ORR） per Investigator assessed using RANO criteria. | 24 Cycles of 28 days each.
Part II (HX301 in combination with temozolomide) :Overall survival（OS） per Investigator assessed using RANO criteria. | 24 Cycles of 28 days each.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital Capital Medical University, Beijing, Beijing Municipality, China